CLINICAL TRIAL: NCT03489798
Title: Comparison of Two Protocols of Misoprostol (PGE1) and Their Effect on the Rate of Cesarean Section Due to Failed Induction. A Randomized, Controlled Trial.
Brief Title: Comparison of Two Protocols of Misoprostol (PGE1) and the Rate of Cesarean Section Due to Failed Induction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Collaborators: Sistema Nacional de Investigadores de Panamá (Unknown)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Investigator - Head: Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2016-04
Record Dates: First submitted 2018-02-13; First posted 2018-04-05 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Induction of Labor
Keywords: Induction of labor; Misoprostol; Failed induction
MeSH Terms: interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 Misoprostol (Experimental): Up to six doses of 25ug of misoprostol applied every 6 hours. End point is cervical Bishop score > 6.
  Interventions: Procedure: 6 misoprostol
- 3 misoprostol (Active Comparator): Up to 3 doses of 25ug of misoprostol applied every 6 hours. End point is cervical Bishop score > 6.
  Interventions: Procedure: 3 misoprostol

INTERVENTIONS:
Procedure: 6 misoprostol — Up to 6 doses of 25ug of misoprostol applied every 6 hours. End point is cervical Bishop score > 6.
  Other Names: Prostaglandin E1 25 ug dose
  Arms: 6 Misoprostol
Procedure: 3 misoprostol — Up to 3 doses of 25ug of misoprostol applied every 6 hours. End point is cervical Bishop score > 6.
  Other Names: Prostaglandin E1 25 ug dose
  Arms: 3 misoprostol

SUMMARY:
To compare two protocols of misoprostol use for cervical ripening: 3 doses (25 ug vaginal each) or up to six doses, every six hours, until an adequate cervical condititon was achieved (BIshop score > 6). In the first group, after 3 doses, the patient was sent to the delivery room for induction with oxytocin and in case of failure, a cesarean section was indicated for this reason. In the second group, up to six doses were used in a similar fashion. Rates of success were evaluated, as well as maternal and fetal complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 34 and 42 weeks of gestation.
* Obstetric indication for termination of pregnancy.
* No fetal evidence of fetal distress

Exclusion Criteria:

* Any contraindication for the use of misoprostol.
* Oligohydramnios.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Vaginal birth | 48 hours
  Number of patients that had a vaginal birth

SECONDARY OUTCOMES:
Maternal complications | 48 hours
  Number of patients that developed a maternal complication due to the use of misoprostol (abruptio placenta, postpartum bleeding, uterine atony).
Fetal complications | 48 hours
  Number of patients that developed a fetal complication due to the use of misoprostol (stillbirth, fetal distress).

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama